CLINICAL TRIAL: NCT02614339
Title: Effect of Adjunctive Metformin on Recurrence of Non-DM Colorectal Cancer Stage II High-risk/ III Colorectal Cancer: Open-label Randomized Controlled
Brief Title: Effect of Adjunctive Metformin on Recurrence of Non-DM Colorectal Cancer Stage II High-risk/ III Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2015-0533
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Non-DM Stage II High-risk Colorectal Cancer; Non-DM Stage III Colorectal Cancer
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Experimental)
  Interventions: Drug: metformin
- control (Active Comparator)
  Interventions: Drug: control

INTERVENTIONS:
Drug: metformin — The patients of this group are treated according to NCCN guideline for stage II high-risk/ III colorectal cancer and receive an additional prescription metformin. Metformin will be prescribed 1g/day (500mg, 2 table/day, or 1000mg, 1 table/day). After adjustment period for 1month, patients who do not have side effects will be taken metformin for additional 47 months (total 48months including the adjustment period).
  Arms: metformin
Drug: control — The patients of this group are treated according to NCCN guideline for stage II high-risk/ III colorectal cancer.
  Arms: control

SUMMARY:
The aim of this study is to identify the effect of adjunctive metformin on recurrence of non-DM Stage II High-risk/ III colorectal cancer. This study is open-label randomized controlled study.

The primary endpoint is to compare the 3-year disease free survival between metformin group and non-metformin group. The secondary endpoint is to compare the 5-year overall survival and disease specific survival between two group, to identify the safety of metformin, and to compare the recurrence rate of polyps after polypectomy between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. patients with stage II high-risk/ III colorectal cancer who were taken an operation for cure, or patients with stage III rectal cancer who were taken an chemoradiation therapy and subsequently operation
2. age 20 - 80 years
3. patients without DM
4. patients who have well performance status for chemotherapy
5. patients who are agreed the study protocol

Exclusion Criteria:

1. patients with DM
2. patients who were diagnosed other cancers (≥ stage II) within 5 years
3. patients who have familial adenomatous polyposis, hereditary non-polyposis colorectal cancer, or inflammatory bowel disease
4. patients who are taken other chemoprevention drugs (ex. NSAIDs, Aspirin)
5. patients who have risk factors to increase lactic acidosis which are renal disease, lung disease, liver disease, or infectious disease
6. Creatinine ≥ 1.5mg/dL (for male), ≥ 1.4mg/dL (for female)
7. patients with congestive heart failure which is needed to treat
8. patients who have allergic history of metformin
9. pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Estimated)
Dates: Start 2015-12; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | after 3 years
  The primary endpoint is to compare 3-year disease free survival between metformin group and non-metformin group.

SECONDARY OUTCOMES:
5-year overall survival | after 5 years
recurrence rate of polyps after polypectomy | after 1 year, and then according to the findings in 1 year colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea